CLINICAL TRIAL: NCT03764319
Title: Low Frequency, Ultra-low Tidal Volume Ventilation in Patients With Severe Acute Respiratory Distress Syndrome and Extracorporeal Membrane Oxygenation: a Prospective, Randomized, Clinical Trial
Brief Title: Low Frequency, Ultra-low Tidal Volume Ventilation in Patients With ARDS and ECMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Martina Hermann, Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MUVienna ARDS-ECMO
Record Dates: First submitted 2018-11-29; First posted 2018-12-05 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2021-09

CONDITIONS: ARDS; Acute Lung Injury; Extracorporeal Membrane Oxygenation; Respiratory Distress Syndrome; Respiratory Tract Diseases; Lung Diseases; Lung Injury, Acute
Keywords: ARDS, ECMO, Ventilation
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome; Respiratory Tract Diseases; Lung Diseases; Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: Comparison of 2 groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Active Comparator): Ultra-protective ventilator settings in patients with ARDS and ECMO.
  Interventions: Other: Ultra-protective ventilator settings
- Control group (Active Comparator): Standard ventilator settings in patients with ARDS and ECMO.
  Interventions: Other: Standard ventilator settings

INTERVENTIONS:
Other: Ultra-protective ventilator settings — 4-5 Breaths per minute; 14-16 cmH2O Positive endexpiratory pressure (PEEP) (adjust PEEP to 23 < Plateau pressure < 25 cmH2O); 23-25 cmH2O Plateau pressure (adjust to not exceed Tidal volume > 4 mL/kg Predicted body weight (PBW)); < 4mL/kg PBW Tidal volume; 1:5 Inspiration:Expiration (I:E)
  Arms: Intervention group
Other: Standard ventilator settings — 12-25 Breaths per minute; 8-12 cmH2O PEEP; max. 35 cmH2O Plateau pressure
  Arms: Control group

SUMMARY:
The acute respiratory distress syndrome (ARDS) is the most severe form of respiratory failure, presented in 10% of all intensive care patients and carrying a high mortality rate. Extracorporeal membrane oxygenation (ECMO) is a rescue treatment for patients with severe ARDS. Mechanical ventilator settings in patients with severe ARDS during ECMO therapy are not clearly defined at the moment.

DETAILED DESCRIPTION:
The aim of this study is to assess the effect of a rigorous low breathing frequency and ultra-low tidal volume ventilation strategy on clinical outcome, compared to standard ventilator settings following the recent guidelines in patients with severe ARDS treated with ECMO.

The hypothesis is that a low breathing frequency and ultra-low tidal volume ventilation strategy is more protective for the ARDS challenged lung and reduces the duration of mechanical ventilation and so increases the ventilator free days in patients with severe ARDS treated with ECMO.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe ARDS - Partial pressure of oxygen/Fraction of inspired oxygen (PaO2/FiO2) < 200 mmHg
* ECMO < 24 hours in situ
* Gender-matched
* Age-matched

Exclusion Criteria:

* BMI > 40
* Expected weaning of ECMO < 3 days (postoperative ECMO)
* Combustion
* Restrictive chest wall impairment
* Pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 44 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Ventilator free days | Immediately after initiation of ECMO up to 28 days
  Ventilator free days
Time from randomization to fulfillment of extubation criteria | Immediately after initiation of ECMO up to 28 days
  Time from randomization (initiation of ECMO) to fulfillment of the extubation criteria:
  * ARDS resolved
  * Temperature ≥ 36°C and ≤ 39°C
  * Low FiO2 (< 0.5)
  * PEEP (< 8 cmH2O) requirement
  * Able to initiate spontaneous breaths
  * Tidalvolume > 5 mL/kg or > 325 mL
  * Minute ventilation 5-6 L/min
  * PaO2/FiO2 > 200 mmHg
  * pH ≥ 7.25
  * Ability to cough after deflating tube cuff
  * Respiratory rate 8-30/min
  * Hemodynamic stability

SECONDARY OUTCOMES:
Total time of mechanical ventilation | Start of mechanical ventilation up to 28 days
  Total time of mechanical ventilation
28 day mortality | Immediately after initiation of ECMO up to 28 days
  Mortality from initiation of ECMO till day 28 after initiation of ECMO
One year mortality | Immediately after initiation of ECMO up to one year
  Mortality from initiation of ECMO till one year after initiation of ECMO
Incidence of reintubation | Immediately after initiation of ECMO up to 28 days
  Incidence of reintubation
Length of ICU stay | Immediately after initiation of ECMO
  Length of ICU stay
Evaluation of RAS, ACE, ACE2. | 2 months
  Analyses of leftover blood. Renin angiotensin system (RAS) and Angiotensin converting enzyme (ACE) evaluation.
Evaluation of Cytokines in pg/ml | 2 months
  IL-6, IL-8, TNFR1, RAGE, Protein C
Evaluation of vitamin D status | Length of ICU stay
  25(OH), 1,25(OH)

CONTACTS AND LOCATIONS:
Overall Officials: Roman Ullrich, Ao.Univ.Prof., Principal Investigator — Department of Anesthesia and Intensive Care
Locations (1):
- Medical University of Vienna - Division of General Anaesthesia and Intensive Care Medicine, Vienna, Austria, Austria